CLINICAL TRIAL: NCT05685069
Title: Prevalence of Attributable Etiology and Modifiable Stroke Risk Factors in Patients With Covert Brain Infarctions (CBI-registry)
Brief Title: Prevalence of Attributable Etiology and Modifiable Stroke Risk Factors in Patients With Covert Brain Infarctions
Acronym: CBI-Registry
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-00293
Record Dates: First submitted 2022-12-21; First posted 2023-01-13 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Silent Stroke; Silent Cerebral Infarct; Covert Brain Infarct; Covert Brain Infarction; Lacune; Silent Brain Infarction
Keywords: Covert brain infarction; Covert cerebrovascular disease; Ischemic stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standardized work-up: A standardized workup procedures including cerebral MRI, long-term rhythm monitoring (3 x 7 days ECG), echocardiography, stroke laboratory, risk factor assessment and noninvasive angiography of the cervical and intracranial arteries will be performed.

SUMMARY:
The CBI registry is a prospective, interdisciplinary, multimodal observational registry of patients with covert brain infarction. Methods: A standardized workup in analogy to manifest ischemic stroke including cerebral MRI, long-term rhythm monitoring (3 x 7 days ECG), echocardiography, laboratory work-up and risk factor assessment as well as noninvasive angiography of the cervical and intracranial arteries will be performed.

DETAILED DESCRIPTION:
Background: Covert brain infarction (CBI) are incidental lesions of presumably vascular etiology, detected on cerebral imaging and without attributable event of an acute ischemic stroke (AIS). Formerly thought to be completely "silent", CBI do have consequences: patients with CBI have a two-fold increased risk of severe stroke in the future, more often covert neurological deficits, and a steeper decline in cognitive function with increased risk of dementia. Important associations of CBI are described with hypertension, carotid stenosis, chronic kidney disease and metabolic syndrome, heart failure, coronary artery disease, hyperhomocysteinemia and obstructive sleep apnea. No trustworthy guidelines exist how to approach a patient with CBI.

Aim and hypothesis: The investigators want to provide a reliable estimate on the yield and relevance of a complete stroke workup to identify modifiable vascular risk factors in patients with CBI searching for an easily treatable cause of the event like a carotid stenosis, atrial fibrillation, hypertension or diabetes. The investigators' hypothesis is that a complete workup in patients with CBI has a similar yield of underlying pathological findings as compared to workup recommended for AIS.

Design: The SILENT registry is a prospective, interdisciplinary, multimodal observational registry of 230 patients with CBI. Methods: A standardized workup procedures including cerebral MRI, long-term rhythm monitoring (3 x 7 days ECG), echocardiography and noninvasive angiography of the cervical and intracranial arteries will be performed.

Statistics: A sample size calculation estimated a sample size of 230 patients. A prespecified analysis protocol will be used.

Significance: This study has the potential to extend the work-up of stroke to patients with CBI. Since CBI are up to three times more frequent than manifest ischemic stroke, this would have huge implications for primary stroke prevention.

ELIGIBILITY:
Inclusion Criteria:

* Any clinically silent ischemic lesions of the brain parenchyma detected on neuroimaging defined according to established criteria as either:

  * DWI positive lesions: Focus of restricted diffusion (high DWI signal and low ADC value) occurring in either white or gray matter, located in the cerebrum, cerebellum, or brain stem AND not satisfying the diagnostic criteria for MS OR
  * Cavitatory Lesions: ≥ 3 mm in size that follow CSF on all sequences that are slit or wedge shaped with an irregular margin AND NOT longitudinally aligned with perforating vessels or with a multiple, bilateral symmetrical distribution OR
  * T2W hyperintense/T1W hypointense lesions: Focal lesion with high T2W signal and low T1W signal that have prior evidence of restricted diffusion; OR present within cortical gray matter or deep gray matter nuclei OR a lesion that is new, compared with an MRI performed within 3 months OR T2W hyper/T1W hypointense lesions in the white matter, which are discontinuous but associated with the classic confluent periventricular T2 intense change of leukoaraiosis (Fazekas ≥2) AND NOT satisfying the diagnostic criteria for MS or with a significant patient history of severe trauma, radiation, drug toxicity, or carbon monoxide poisoning
* Informed Consent as documented by signature by patient or legally authorized representative

Exclusion Criteria:

* Projected life expectancy of less than 2 years,
* Contraindication to MRI,
* Patients with a history of symptoms compatible with an AIS/TIA attributable to the lesion observed, covert neurological deficits are allowed,
* Patient is already included in another clinical trial that will affect the objectives of this study,
* Patient's lack of accountability, inability to appreciate the nature, meaning and consequences of the study and to formulate his/her own wishes correspondingly,
* Women who are pregnant or breast feeding or intention to become pregnant during the course of the study,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Contraindications to any of the routine procedures, e.g. inability to obtain neurovascular ultrasound examination,
* Known or suspected non-compliance, drug or alcohol abuse

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited by the Neuroradiology Department of Inselspital Bern. All patients undergoing a brain MRI showing a presumably silent brain lesion and fulfilling the inclusion/exclusion criteria will be eligible for the study. Inpatients will be contacted while on a ward and outpatients by telephone calls.
Sampling Method: Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Modified Trial of Org 10172 in Acute Stroke Treatment etiology | After baseline work-up, expected to be at least 3 months after brain imaging
  Incorporating results from the baseline work-up the most likely etiology according to the modified Trial of Org 10172 in Acute Stroke Treatment (TOAST) for the chronic brain lesions observed will be rated:
  * Large vessel atherothrombotic stroke: >=50% ipsilateral vascular stenosis present
  * Cardiac embolism: Sustained or paroxysmal atrial fibrillation or atrial flutter and/or Structural or functional high-risk source of embolism
  * Small vessel (lacunar) stroke: ischemia in perforating brain artery without embolic source
  * Patent foramen ovale (PFO): PFO with or without atrial septal aneurysm with recommendation for closure (patient age <60 OR patient age 60-70 and Risk of Paradoxical Embolism (RoPE) Score ≥5
  * Other specific etiology (e.g. dissections)
  * Stroke of undetermined etiology (two or more causes identified, negative evaluation)

SECONDARY OUTCOMES:
Percentage of Modified Trial of Org 10172 in Acute Stroke Treatment etiology | At the end of follow-up (2 years)
  Incorporating results from the baseline work-up the most likely etiology according to the modified Trial of Org 10172 in Acute Stroke Treatment (TOAST) for the chronic brain lesions observed will be rated:
  * Large vessel atherothrombotic stroke: >=50% ipsilateral vascular stenosis present
  * Cardiac embolism: Sustained or paroxysmal atrial fibrillation or atrial flutter and/or Structural or functional high-risk source of embolism
  * Small vessel (lacunar) stroke: ischemia in perforating brain artery without embolic source
  * Patent foramen ovale (PFO): PFO with or without atrial septal aneurysm with recommendation for closure (patient age <60 OR patient age 60-70 and Risk of Paradoxical Embolism (RoPE) Score ≥5
  * Other specific etiology (e.g. dissections)
  * Stroke of undetermined etiology (two or more causes identified, negative evaluation)
Median of National Institute of Health Stroke score (NIHSS) | At baseline visit, expected to be at least 3 months after brain imaging
  The NIHSS is a 15-item neurological examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. A trained observer rates the patent's ability to answer questions and perform activities, without coaching and without making assumptions about what the patient can do.
  Ratings for each item are scored on a 3- to 5-point scale, with 0 as normal, and there is an allowance for untestable items. Scores range from 0 to 42, with higher scores indicating greater severity.
Percentage of Presence of covert neurological deficits corresponding to the CBI | At baseline visit, expected to be at least 3 months after brain imaging
  Unrecognized or unreported stroke-like symptoms, called covert symptoms, e.g. visual field defect or slight ataxia
Median of Modified Rankin Scale functional status (mRS) | At baseline visit, expected to be at least 3 months after brain imaging
  The Modified Rankin Scale (mRS) assesses disability in patients who have suffered a stroke and is compared over time to check for recovery and degree of continued disability. A score of 0 is no disability, 5 is disability requiring constant care for all needs; 6 is death.
Median of Montreal Cognitive Assessment (MOCA) | At baseline visit, expected to be at least 3 months after brain imaging
  The Montreal Cognitive Assessment (MoCA) was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The MoCA may be administered by anyone who understands and follows the instructions, however, only a health professional with expertise in the cognitive field may interpret the results. Time to administer the MoCA is approximately 10 minutes. The total possible score is 30 points; a score of 26 or above is considered normal.
Median of Becks-Depression-Inventar-II | At baseline visit, expected to be at least 3 months after brain imaging
  The Beck Depression Inventory (BDI, BDI-1A, BDI-II), created by Aaron T. Beck, is a 21-question multiple-choice self-report inventory. Like the BDI, the BDI-II also contains about 21 questions, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms. The standardized cutoffs used differ from the original:
  0-13: minimal depression 14-19: mild depression 20-28: moderate depression 29-63: severe depression.
Median of EuroQol-5d | At baseline visit, expected to be at least 3 months after brain imaging
  The EQ-5D consists of several components: On the one hand, the self-assessment using the EQ-5D questionnaire, which describes the state of health using five dimensions:
  Agility, mobility the ability to take care of yourself Everyday activities (e.g. work, studies, housework, family, free time) pain, physical discomfort fear, depression
Number of Participants with Dyslipidemia | After baseline work-up, expected to be at least 3 months after brain imaging
  according to the 2018 ACC/AHA recommendations
Number of Participants with New diagnosis of diabetes mellitus type 2 | After baseline work-up, expected to be at least 3 months after brain imaging
  Elevated HbA1c or random glucose according to the 2017 International Diabetes Federation Guidelines
Number of Participants with Hematological abnormality | After baseline work-up, expected to be at least 3 months after brain imaging
  requiring change of management
Number of Participants with Abnormality in renal function or electrolytes | After baseline work-up, expected to be at least 3 months after brain imaging
  requiring change of management
Number of Participants with Ischemic stroke | At the end of follow-up (2 years)
  defined as new sudden focal neurological deficit of presumed cerebrovascular etiology, occurring > 24 hours after the index SBI, that persisted beyond 24 hours and was not due to another identifiable cause
Number of Participants with TIA | At the end of follow-up (2 years)
  defined as a transient episode of neurologic dysfunction caused by focal brain, spinal cord, or retinal ischemia without cerebral infarction on imaging
Number of Participants with Myocardial infarction | At the end of follow-up (2 years)
  defined as typical symptoms and cardiac biomarker elevation (troponin I or T, creatine kinase-MB) above the upper limit of normal, new pathological Q waves in at least 2 contiguous electrocardiogram leads, or confirmation at autopsy or by coronary angiography or by MRI.
Number of Participants with relevant symptomatic intracranial hemorrhage | At the end of follow-up (2 years)
  including subdural, epidural, subarachnoidal and intracerebral hemorrhage, defined as hemorrhage that leads to a clinical worsening and hospitalisation and is assessed by the treating physician to be likely the cause of the new neurological symptom or the death. Intracerebral hemorrhage due to a trauma will not be considered.
Number of Participants with Major cardiovascular events | At the end of follow-up (2 years)
  defined as composite of stroke, myocardial infarct, heart failure or cardiovascular death)
Number of Participants with Systemic embolism | At the end of follow-up (2 years)
  defined as abrupt vascular insufficiency associated with clinical or radiological evidence of arterial occlusion of an extremity or organ in absence of another likely mechanism (e.g. atherosclerosis, instrumentation or trauma)
Number of Participants with Vascular death | At the end of follow-up (2 years)
  defined as death that is due to a vascular cause
Number of Participants with All-cause mortality | At the end of follow-up (2 years)
  defined as death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Urs Fischer, Prof. Dr. med., Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (2):
- Centre Hospitalier Universitaire de Tours, Tours, France
- Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Open to expand the registry to other centers. Can provide the materials:
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: From 2022 onwards
Access Criteria: After clearance by ethics

REFERENCES:
- [Background] Meinel TR, Kaesmacher J, Roten L, Fischer U. Covert Brain Infarction: Towards Precision Medicine in Research, Diagnosis, and Therapy for a Silent Pandemic. Stroke. 2020 Aug;51(8):2597-2606. doi: 10.1161/STROKEAHA.120.030686. Epub 2020 Jul 10. No abstract available. PMID 32646332
- See also: Substudy offering implantable cardiac monitors to patients with CBI and high risk for atrial fibrillation — https://clinicaltrials.gov/ct2/show/NCT04449523